CLINICAL TRIAL: NCT04091750
Title: Phase II Study of Nivolumab/Ipilimumab Plus Cabozantinib in Patients With Unresectable Advanced Melanoma
Brief Title: Nivolumab/Ipilimumab Plus Cabozantinib in Patients With Unresectable Advanced Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: MedStar Franklin Square Medical Center (Other); Hackensack Meridian Health (Other); Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000904
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Melanoma
Keywords: melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Nivolumab 3mg/kg IV plus Ipilimumab 1mg/kg IV every 3 weeks x 4 cycles with Cabozantinib 40mg PO daily for 12 weeks (Induction); Followed by Maintenance therapy: Nivolumab 480mg IV every 4 weeks for up to 92 weeks; Cabozantinib 40mg PO daily for up to 92 weeks; Maintenance therapy will continue for up to 92 weeks to complete 2 years total of treatment if tolerating therapy well and disease is controlled.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Cabozantinib

INTERVENTIONS:
Drug: Nivolumab — Induction: 3mg/kg IV every 3 weeks x 4 cycles
  Maintenance: 480mg IV every 4 weeks for up to 92 weeks
  Other Names: Opdivo
Drug: Ipilimumab — Induction: 1mg/kg IV every 3 weeks x 4 cycles
  Other Names: Yervoy
Drug: Cabozantinib — Induction and Maintenance: 40mg PO daily
  Other Names: Cabometyx

SUMMARY:
In this phase II advanced melanoma study, all patients will receive treatment with nivolumab/ipilimumab plus cabozantinib for a 12 week induction period followed by nivolumab plus cabozantinib maintanence to complete up to 2 years of therapy unless disease progression, dose limiting toxicity, provider/patient decision or patient withdrawal of consent occurs. The primary endpoint is the one year PFS rate. Patients will have staging scans at baseline and every 12 weeks during the first 2 years on study. Safety evaluations including labs, EKG and history and physical will occur at each visit. Baseline tumor sample is required and on treatment biopsy will be optional of superficial tumor in the skin, subcutaneous tissue or lymph node that is palpable.

DETAILED DESCRIPTION:
Subjects will receive nivolumab, ipilimumab and cabozantinib until either disease progression, the occurrence of unacceptable drug-related toxicity or for other reason(s) for subject withdrawal. Treatment will continue for up to 2 years unless there is disease progression, drug intolerance or other reason for discontinuation discussed with the principal investigator (PI). Patients with ongoing complete or partial response may discontinue therapy after 1 year on treatment at the discretion of the treating investigator.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have unresectable stage IIIb-IIId or IV melanoma by AJCC 8th edition. Note: Patients with uveal melanoma are excluded from this study.
2. Age > 18 and ECOG Performance Status of 0 or 1.
3. Measurable disease by RECIST 1.1
4. Baseline tumor specimen available.
5. Recovery to baseline or ≤ Grade 1 CTCAE v4 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
6. Adequate organ and marrow function.
7. Capable of understanding and complying with the protocol requirements and must have signed the informed consent document.
8. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment.
9. Female subjects of childbearing potential must not be pregnant at screening.

Exclusion Criteria:

1. Prior treatment with anti-PD-1/PD-L1 therapy, anti-CTLA-4 therapy or cabozantinib. Prior adjuvant anti-PD-1 and/or anti-CTLA-4 therapy is allowed if relapse is greater than 6 months from last dose.
2. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment.
3. Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment.
4. Radiation therapy for bone metastasis or brain metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before the first dose of study treatment.
5. Known brain metastases that are >10mm or cranial epidural disease unless adequately treated with radiosurgery and/or surgery (including radiosurgery). Eligible subjects must be neurologically asymptomatic and without corticosteroid requirement. Dexamethasone < 2mg daily (or equivalent) will be allowed if discontinuation of corticosteroids is not feasible due to post-radiation effects and patient is asymptomatic. Patients with active, asymptomatic brain metastases that are <10mm and no corticosteroid requirement will be allowed without radiosurgery or surgery.
6. History of active autoimmune disorder requiring immunosuppressive agents. Patients with autoimmune disorders considered low risk, such as vitiligo and thyroiditis, will be allowed.
7. Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g. dabigatran), betrixaban, or platelet inhibitors (eg, clopidogrel).

   Allowed anticoagulants are the following:
   1. Prophylactic use of Low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH) are permitted.
   2. Anticoagulation with therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban is allowed in subjects without known brain metastases who are on a stable dose of LMWH anticoagulant for at least 6 weeks 1week before first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
8. The subject has prothrombin time (PT)/INR or partial thromboplastin time (PTT) test ≥ 1.3 x the laboratory ULN within 7 days before the first dose of study treatment.
9. The subject has uncontrolled, significant intercurrent or recent illness.
10. Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks before first dose of study treatment.
11. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 28 days before first dose of study treatment.
12. Pregnant or lactating females.
13. Inability to swallow tablets.
14. Previously identified allergy or hypersensitivity to components of the study treatment formulations.
15. Diagnosis of another malignancy within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy.
16. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey T Gibney, MD, Principal Investigator — MedStar Georgetown University Hospital
Locations (3):
- United States (3):
  - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Medstar Franklin Square Medical Center, Harry and Jeanette Weinberg Cancer Institute, Baltimore, Maryland
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Induction phase:
  Nivolumab 3mg/kg IV plus Ipilimumab 1mg/kg IV every 3 weeks x 4 cycles (12 week period)
  Cabozantinib 40mg PO daily for 12 weeks
  Maintenance phase:
  Nivolumab 480mg IV every 4 weeks for up to 92 weeks
  Cabozantinib 40mg PO daily for up to 92 weeks
  Maintenance therapy will continue for up to 92 weeks to complete 2 years total of treatment if tolerating therapy well and disease is controlled.
  Nivolumab: Induction: 3mg/kg IV every 3 weeks x 4 cycles
  Maintenance: 480mg IV every 4 weeks for up to 92 weeks
  Ipilimumab: Induction: 1mg/kg IV every 3 weeks x 4 cycles
  Cabozantinib: Induction and Maintenance: 40mg PO daily
Period: Overall Study
Arm/Group | Single Arm
Started | 14
Completed | 9
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: The Progression Free Survival (PFS) for Nivolumab/Ipilimumab Plus Cabozantinib in Patients With Unresectable Advanced Melanoma.
Description: The PFS rate for nivolumab/ipilimumab plus cabozantinib in patients with unresectable advanced melanoma using imRECIST.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 14
Participants | 6

2. Secondary Outcome: The Response Rate of Nivolumab/Ipilimumab Plus Cabozantinib in Patients With Unresectable Advanced Melanoma.
Description: The ORR by imRECIST of nivolumab/ipilimumab plus cabozantinib in patients with unresectable advanced melanoma.
Time Frame: 1 year
Reporting Status: Not Posted

3. Secondary Outcome: The Overall Survival (OS) of Patients With Unresectable Advanced Melanoma Treated With Nivolumab/Ipilimumab Plus Cabozantinib.
Description: The median and 3 year OS rate of patients with unresectable advanced melanoma treated with nivolumab/ipilimumab plus cabozantinib.
Time Frame: 3 years
Reporting Status: Not Posted

4. Secondary Outcome: The Incidence of Treatment-emergent Adverse Events of Nivolumab/Ipilimumab Plus Cabozantinib in Patients With Unresectable Advanced Melanoma.
Description: The rate of all grade and grade 3-5 adverse events and the rate of discontinuation of study drug(s) due to adverse events.
Time Frame: 2 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Associations Between Baseline Tumor Mutational Burden (TMB), Angiogenesis Pathways, and Immunophenotyping With Clinical Activity of Nivolumab/Ipilimumab Plus Cabozantinib in Patients With Unresectable Advanced Melanoma.
Description: Measured in terms of ORR, PFS, and OS.
Time Frame: 3 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Associations Between Baseline Mutations in Genes Regulating Anti-tumor Immunity With Tumor Immunophenotype and Clinical Activity of Nivolumab/Ipilimumab Plus Cabozantinib in Patients With Unresectable Advanced Melanoma.
Description: Measured in terms of ORR, PFS, and OS.
Time Frame: 3 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: On Treatment Biopsy for Evidence of Increased Immune Infiltration, Vascularization, and MHC Expression to Nivolumab/Ipilimumab Plus Cabozantinib in Patients With Unresectable Advanced Melanoma.
Description: Measured by the change in immune cell populations, CD31 vascularization, and MHC class I expression by multiplex immunofluorescense (IF) between baseline and on treatment tumor specimens.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from after informed consent through 30 days after the decision to discontinue study treatment (approximately 2 years); All Cause Mortality was collected after discontinuation of treatment until death during a long term follow up period (approximately 4 years).
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 10/14
Serious Adverse Events (participants affected / at risk) | 9/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=14)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Double vision
Abdominal pain (Gastrointestinal disorders) | 1 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 2 (3)
Non-cardiac chest pain (General disorders) | 1 (2)
Catheter related infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=14)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) — Thyroiditis
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypoparathyroidism (Endocrine disorders) | 1 (1)
Hypophysitis (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (1) — left eye swelling
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Dry eyes
Eye disorders - Other, specify (Eye disorders) | 1 (1) — itchy eye (left)
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Flashing lights/white circles
Eye disorders - Other, specify (Eye disorders) | 1 (1) — itchiness both eyes
Watering eyes (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (8)
Belching (Gastrointestinal disorders) | 1 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 6 (22)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Enterocolitis (Gastrointestinal disorders) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (4)
Mucositis oral (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (5)
Oral pain (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 3 (10)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 3 (4)
Fatigue (General disorders) | 6 (9)
Fever (General disorders) | 3 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — vision changes
Pain (General disorders) | 3 (3)
Allergic reaction (Immune system disorders) | 2 (2)
Bronchial infection (Infections and infestations) | 2 (2)
Paronychia (Immune system disorders) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (5)
Wound infection (Infections and infestations) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 8 (16)
Alkaline phosphatase increased (Investigations) | 3 (6)
Aspartate aminotransferase increased (Investigations) | 8 (18)
CPK increased (Investigations) | 2 (21)
Creatinine increased (Investigations) | 5 (7)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
GGT increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 2 (6)
Neutrophil count decreased (Investigations) | 1 (1)
Serum amylase increased (Investigations) | 3 (4)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 3 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (15)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) — lactic acidosis
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dysesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (6)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Irritability (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (6)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Renal calculi (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 (15)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (6)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (4)
Hypotension (Vascular disorders) | 2 (2)
Phlebitis (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Vascular disorder- Other, specify (Vascular disorders) | 1 (1) — carotid artery blockage
Vascular disorder- other, specify (Vascular disorders) | 1 (1) — popliteal artery blockage

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT04091750/Prot_SAP_000.pdf